CLINICAL TRIAL: NCT06707844
Title: Comparison of Tissue Flossing and Myofascial Release on Calf Muscles in Patients With Pes Planus
Brief Title: TF and MFR on Calf Muscles in Patients With Pes Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/MS-PT/02019 Arfa Zafar
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Pes Planus
Keywords: tissue flossing; Flatfeet; myofascial release; balance; arch height; range of motion
MeSH Terms: conditions — Flatfoot | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tissue flossing (Experimental): * Tissue flossing involves wrapping a latex band around the calf muscles with 50-75% elongation, followed by active ankle movements (dorsiflexion, plantarflexion, circles, heel raises).
  * Protocol: 4 sets of 8 repetitions, 10-second rest between sets
  * Performed twice weekly for 3 weeks.
  Conventional Treatment
  Interventions: Other: Conventional treatment; Other: Tissue flossing
- Myofascial release (Active Comparator): * Myofascial release is a manual therapy applying sustained pressure on the calf muscles to release fascial restrictions.
  * Protocol: 3 sets of 2-minute pressure applications with a 1-minute break between sets
  * Performed twice weekly for 3 weeks
  Conventional Treatment
  Interventions: Other: Conventional treatment; Other: Myofascial release

INTERVENTIONS:
Other: Conventional treatment — Conventional treatment will include:
  * Stretching exercises (5Reps with 15sec hold): Gastrocnemius-soleus stretch, TA stretch.
  * Strengthening exercises (5Sets, 5Reps, 5sec hold): Weight-bearing lunges, Short-foot exercise.
  * Maitland mobilization Grade 2 & 3 (3 Sets, 20Reps) at Talonavicular joint.
Other: Myofascial release — * Myofascial release is a manual therapy applying sustained pressure on the calf muscles to release fascial restrictions.
  * Protocol: 3 sets of 2-minute pressure applications with a 1-minute break between sets
  * Performed twice weekly for 3 weeks
  Arms: Myofascial release
Other: Tissue flossing — Tissue flossing involves wrapping a latex band around the calf muscles with 50-75% elongation, followed by active ankle movements (dorsiflexion, plantarflexion, circles, heel raises).
  Protocol: 4 sets of 8 repetitions, 10-second rest between sets Performed twice weekly for 3 weeks.
  Arms: Tissue flossing

SUMMARY:
Pes planus, commonly known as flat feet, is a condition characterized by a reduced or absent arch in the foot, which often leads to pain and functional limitations. This study aims to evaluate the effectiveness of two therapeutic interventions-tissue flossing and myofascial release-in improving balance, arch height, and range of motion (ROM) in patients with flexible flatfoot. The research will be conducted at the Margalla Rehabilitation Center over a duration of six months, involving a total of 44 participants divided into two equal groups. One group will receive tissue flossing as the intervention, while the other group will undergo myofascial release. Participants will be selected using non-probability convenience sampling. Eligible individuals will be adults aged 18-25 years with flexible pes planus and limited ankle dorsiflexion. The study seeks to provide valuable insights into the comparative effectiveness of these interventions for managing symptoms associated with flat feet. Data was be analyzed through SPSS version 25.

DETAILED DESCRIPTION:
Pes planus, or flat feet, is characterized by a reduced or absent arch, causing the entire sole to contact the ground. It is categorized into flexible and rigid types, with flexible pes planus being more common. In this form, the arch is visible in non-weight-bearing positions but flattens during standing or walking, while rigid pes planus remains flat irrespective of weight-bearing. The condition often results in foot instability, excessive eversion, and midfoot abduction, leading to pain, fatigue, and reduced shock absorption during activities.

Flexible flatfoot is prevalent in children but can persist into adulthood, affecting 2% to 23% of adults in the U.S. and 13.6% in India. It disrupts gait mechanics, shifting weight medially, impairing balance, and increasing injury risk. Management ranges from conservative treatments like physical therapy to surgical interventions in severe cases.

Emerging therapies include tissue flossing and myofascial release (MFR). Tissue flossing uses compression bands to improve blood flow, reduce pain, and enhance range of motion (ROM). In contrast, MFR applies sustained pressure to relieve fascial tension, promoting flexibility and reducing discomfort. Both techniques show promise for addressing the biomechanical and functional impairments associated with pes planus.

Literature review: According to literature, Galis et al. (2022) performed a study that aimed to examine the effects of applying tissue flossing band at different pressure levels on ankle ROM, strength and power performance in university students. The results showed an increase in dorsiflexion ROM and power. Furthermore, the author concluded that this can aid injury prevention, performance enhancement, and functional ability.

In another study, Driller et al. (2016) conducted a study on the effects of tissue flossing on ankle ROM and jump performance in recreational athletes. The study concluded that applying floss bands to the ankle effectively increased both dorsiflexion and plantarflexion ROM and enhances single-leg jump performance in recreational athletes.

Similarly, Choi et al. (2022) conducted a study aimed at investigating the impact of myofascial release of the peroneus longus muscle on the activity of the abductor hallucis muscle and the medial longitudinal arch in individuals with flexible pes planus. The results showed an increase in abductor hallucis muscle activity and elevation of the medial longitudinal arch.

A study conducted by Chang et al. (2021) examined the effect of a single session of tissue flossing on the knee joint in female college students. The results showed a significant improvement with a medium-to-large effect in the Y-Balance test assessment immediately postintervention. He concluded that tissue flossing can indeed enhance dynamic balance.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-25 years.
* Having normal BMI ranging from 18.5 to 24.9 kg/m²
* Having flexible flat feet, defined as a navicular drop test value of ≥10 mm
* Must have pain in the calf muscles or ankle joint, with a NPRS score of ≥3
* Must have limited ankle dorsiflexion ROM, defined as ≤10° of dorsiflexion

Exclusion Criteria:

* Patients with rigid flatfoot
* History of ankle or calf muscle injury or surgery within the last 6 months
* Individuals with latex allergy
* Individuals having any lumbo-pelvic, hip, knee and ankle pathologies such as fractures, dislocations, degenerative diseases etc.
* Any neurological disease
* Pregnant females
* Individuals with BMI greater than or equal to 25.0 kg/m²
* Ongoing use of medications such as muscle relaxants or anti-inflammatory drugs
* Involved in athletic training

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-01-21 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 3 weeks
  This tool will be used to assess pain intensity, at baseline, 2nd week and 3rd week post treatment

SECONDARY OUTCOMES:
Digital Goniometer | 3 weeks
  It will be used for the measurement of ankle range of motion. Changes from baseline, 2nd week and 3rd week will be taken.
Brody's Navicular Drop Test | 3 weeks
  It will be used for the measurement of navicular drop. It is the one of the static foot assessment tools and is intended to represent the displacement of the navicular tuberosity from a neutral position. Measurements taken at baseline, 2nd week and 3rd week
Single-Leg Stance Test | 3 weeks
  It will be used to assess each patient's static balance with their eyes open and arms on hips. Good static balance is indicated by participant's ability to maintain position for atleast 30 seconds. Test will be repeated 3 times and average will be taken. measurements will be taken at baseline, 2nd week and 3rd week.
Y-Balance test | 3 weeks
  It will be used for dynamic balance assessment. Patient is asked to stand on one leg while reaching out in 3 different directions (anterior, posteromedial and posterolateral) with the other lower extremity.

CONTACTS AND LOCATIONS:
Overall Officials: Aneela Zia, MsOMPT, Principal Investigator — Riphah International University
Locations (1):
- Margalla Rehabilitation Center, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. R A, Malar A, J H, G S. The cause and frequency of PES Planus (Flat Foot) problems among young adults. Asian Journal of Medical Sciences. 2021;12(7):107-11.